CLINICAL TRIAL: NCT01089777
Title: Monitoring and Characterization of Coronary Flow By Transthoracic Parametric Doppler (TPD) During Exercise Stress Test
Status: Terminated | Type: Observational
Sponsor: Echosense Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DOP04
Record Dates: First submitted 2010-03-16; First posted 2010-03-19 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2011-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ultrasound Doppler monitoring — Ultrasound Doppler monitoring throughout the stress test

SUMMARY:
The study is an open prospective study of coronary flow preferably of the left anterior descending artery (LAD), by a Transthoracic Parametric Doppler (TPD) system during conventional exercise stress test. The system is a noninvasive non-imaging device designed to monitor coronary flow velocity and display the data continuously during exercise stress tests. The system enables continuous monitoring of coronary flow during resting, stress loading and recovery phases. The study intent is to improve the stress test predictive value for CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Planned for ergometry test
* Signed informed consent

Exclusion Criteria:

* Excluded for stress test on a treadmill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scheduled to exercise stress test
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Monitor coronary artery flow during exercise stress test. | 1-3 months following the stress test

SECONDARY OUTCOMES:
Improve CAD predictive power of stress testing | 1-3 months following the stress test

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular department, Carmel medical center, Haifa, Israel